CLINICAL TRIAL: NCT01464034
Title: A Multi-Center Phase I/II, Open-Label, Dose-Finding Pilot Study of the Combination of Carfilzomib and Pomalidomide With Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Safety and Efficacy Study of Carfilzomib and Pomalidomide With Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Criterium, Inc. (Industry)
Collaborators: Amgen (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMyC 10-MM-01; IST-CAR-521 (Other: Onyx Pharmaceuticals); PO-MM-PI-0034 (Other: Celgene Corporation)
Record Dates: First submitted 2011-10-19; First posted 2011-11-03 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; pomalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib, Pomalidomide, Dexamethasone (Experimental): All eligible subjects will receive the study intervention of Carfilzomib, Pomalidomide, and Dexamethasone.
  Interventions: Drug: Carfilzomib; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — IV over 30 minutes on Days 1,2,8,9,15, and 16 every 28 days
  Other Names: PR-171
Drug: Pomalidomide — PO daily on Days 1-21, every 28 Days
  Other Names: CC-4047
Drug: Dexamethasone — 40 mg weekly PO or IV on Days 1, 8, 15, and 22, every 28 days.
  Other Names: Decadron

SUMMARY:
This is a dose finding pilot study to evaluate the safety and determine the maximum tolerated dose of the combination of carfilzomib and pomalidomide with dexamethasone (CPD) in patients with relapsed or refractory multiple myeloma followed by a phase II expansion at the MTD to evaluate efficacy.

DETAILED DESCRIPTION:
This is a dose finding pilot study to evaluate the safety and determine the maximum tolerated dose of the combination of carfilzomib and pomalidomide with dexamethasone (CPD) in patients with relapsed or refractory multiple myeloma followed by a phase II expansion at the MTD to evaluate efficacy. The study will explore the efficacy of CPD including overall response, time to progression, progression free survival, and time to next therapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytopathologically or histologically confirmed dx of multiple myeloma
* Relapsed or refractory to the most recently received therapy.
* All pts must have received prior lenalidomide therapy and been determined to be refractory, relapsed, or intolerant.
* Measurable disease, as indicated by one or more of the following:

Serum M-protein ≥ 0.5 g/dL Urine Bence Jones protein ≥ 200 mg/24 hr Elevated Free Light Chain as per IMWG criteria, and abnormal ratio

* Pts must be ≥ 18 years of age
* Life expectancy of more than 3 months
* ECOG PS of 0-2
* Adequate hepatic function, with bilirubin < 2 times the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times ULN
* Uric acid must be within laboratory normal range
* CrCl ≥ 50 mL/min
* Additional Laboratory Requirements ANC ≥1.0 x 109/L Hgb ≥8 g/dL(transfusion permitted) Platelet count ≥50.0 x 109/L
* Screening ANC should be independent of granulocyte-and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for at least 2 weeks
* Pts may receive RBC or platelet transfusions, if clinically indicated, in accordance with institutional guidelines
* Screening platelet count should be independent of platelet transfusions for at least 2 weeks.
* Written informed consent in accordance with federal, local, and institutional guidelines
* FCBP must agree to ongoing pregnancy testing
* FCBP must have a negative serum or urine pregnancy test and agree to birth control.
* Male pts must agree to never have unprotected sexual contact with a female who can become pregnant and must agree to either completely abstain from sexual contact with females who are pregnant or are able to become pregnant. The patient must agree to inform his physician if he has had unprotected sexual contact with a female who can become pregnant or if he thinks for any reason that his sexual partner may be pregnant.
* Male pts cannot donate semen or sperm while taking pomalidomide and for 28 days after completing the study.
* All pts must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Pts must agree to take enteric-coated aspirin 81 mg orally daily, or if history of prior thrombotic disease, must be fully anticoagulated with warfarin (INR 2-3) or be treated with full-dose, low molecular weight heparin, as if to treat deep venous thrombosis (DVT)/pulmonary embolism (PE)at the investigator's discretion

Exclusion Criteria:

* Pts with known sensitivity to any immunomodulatory drugs (IMiDs)
* Use of any other experimental drug or therapy within 21 days prior to first dose
* Exposure to any prior chemotherapy, steroid use, or other myeloma treatment within 14 days prior to first dose. Pts currently on long term steroids do not require any washout period. in addition, steroid use for spinal cord compression is permitted and does not require a washout period.
* Radiation therapy within 14 days prior to first dose
* Known allergies to carfilzomib or Captisol
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Current diagnosis of plasma cell leukemia
* Waldenström's macroglobulinemia
* Major surgery within 21 days prior to first dose
* Pregnant or lactating females
* Congestive heart failure (NYHA class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction in the previous six months prior to first dose.
* Uncontrolled hypertension
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within 14 days prior to first dose
* Pts receiving active treatment or intervention for any other malignancy or pts who, at the Investigator's discretion, may require active treatment or intervention for any other malignancy within 8 months of starting study treatment.
* Serious psychiatric or medical conditions that could interfere with treatment
* Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose and/or within 14 days before enrollment
* Contraindication to any of the required concomitant drugs, including proton-pump inhibitor (e.g. lansoprazole), enteric-coated aspirin or if a history of prior thrombotic disease, warfarin or low molecular weight heparin
* Pts in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g. due to pre-existing pulmonary, cardiac, or renal impairment
* Pts with primary systemic amyloidosis
* Pts who have received prior treatment with carfilzomib (Phase II only)
* Pts who have received prior treatment with pomalidomide (Phase II only)
* Pts who have received prior treatment with both carfilzomib & pomalidomide (Phase I only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2011-11; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events as a Measure of Safety and Tolerability | Throughout treatment, estimated at 2-12 months per patient
  Review of adverse events for safety and to determine the maximum tolerated dose of the combination treatment.
Overall Response in Phase II | Every 28 days while on treatment (estimated at 2- 12 months per patient)
  Overall Response (SD, MR, PR, VGPR, CR, sCR)

SECONDARY OUTCOMES:
Overall Response in Phase I | Every 28 days while on treatment (estimated at 2- 12 months per patient)
  Overall response (SD, MR, PR, VGPR, CR, sCR)
Time to Progression | Every 28 days while on treatment (estimated at 2-12 months per patient)
Progression Free Survival | throughout follow up (every 2-3 months for 2 years)
Time to next therapy | throughout follow up (every 2-3 months for 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Jatin Shah, MD, Principal Investigator — AMyC; Brian GM Durie, MD, Principal Investigator — AMyC
Locations (9):
- United States (9):
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - The John Theurer Cancer Center @ Hackensack UMC, Hackensack, New Jersey
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Shah JJ, Stadtmauer EA, Abonour R, Cohen AD, Bensinger WI, Gasparetto C, Kaufman JL, Lentzsch S, Vogl DT, Gomes CL, Pascucci N, Smith DD, Orlowski RZ, Durie BG. Carfilzomib, pomalidomide, and dexamethasone for relapsed or refractory myeloma. Blood. 2015 Nov 12;126(20):2284-90. doi: 10.1182/blood-2015-05-643320. Epub 2015 Sep 17. PMID 26384354